CLINICAL TRIAL: NCT05488587
Title: Serum Levels of Some Trace Elements in Hepatocellular Carcinoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Atef Fadel Ibrahem, Resident at Tropical Medicine and Gastroenterology, Sohag University
Other Study IDs: Soh-Med-22-07-11
Record Dates: First submitted 2022-07-19; First posted 2022-08-04 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- hepatocellular carcinoma
  Interventions: Diagnostic Test: magnesium and zinc levels
- liver cirrhosis
  Interventions: Diagnostic Test: magnesium and zinc levels
- healthy individuals
  Interventions: Diagnostic Test: magnesium and zinc levels

INTERVENTIONS:
Diagnostic Test: magnesium and zinc levels — measuring magnesium and zinc levels

SUMMARY:
Hepatocellular carcinoma (HCC) is the sixth most frequent malignancy worldwide, with an estimated 906,000 new cases and 830,000 deaths in 2020. It is also the third leading cause for cancer deaths, with 15% 5-year survival rate .

Diagnosis of HCC in cirrhotic patients is mainly based on non-invasive imaging techniques. Multiphasic computed tomography (CT) and dynamic contrast-enhanced magnetic resonance imaging (MRI) are the most sensitive imaging techniques for diagnosis of HCC. While the most common serologic marker for early screening of HCC is alpha-fetoprotein (AFP) .

Liver is the main site of trace elements metabolism, and their levels are affected by different causes of liver disease .

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the sixth most frequent malignancy worldwide, with an estimated 906,000 new cases and 830,000 deaths in 2020. It is also the third leading cause for cancer deaths , with 15% 5-year survival rate.

Diagnosis of HCC in cirrhotic patients is mainly based on non-invasive imaging techniques. Multiphasic computed tomography (CT) and dynamic contrast-enhanced magnetic resonance imaging (MRI) are the most sensitive imaging techniques for diagnosis of HCC. While the most common serologic marker for early screening of HCC is alpha-fetoprotein (AFP).

Liver is the main site of trace elements metabolism, and their levels are affected by different causes of liver disease. Zinc (Zn) is an essential trace element which is required for the function of numerous enzymatic molecules active in human cell metabolic pathways. Zn plays an important role in cell growth, differentiation, apoptosis, and metabolism, with more than 300 proteins that regulate cellular functions containing Zn-binding domains. Zn protects against carcinogenesis as it helps activation of deoxyribonucleic acid (DNA) repair enzymes. Also it is a component of superoxide dismutase, an enzyme that removes free radicals.

Zn deficiency was reported to be associated with increased liver fibrosis.and hepatitis C virus (HCV) related HCC. Zn deficiency is also associated with complications related to liver cirrhosis, such as sarcopenia and hepatic encephalopathy.

Magnesium (Mg), as a co-factor for up to 600 enzymes, has a fundamental role in many physiological and biochemical functions including cell proliferation, DNA repair and energy metabolism.

The available data indicate an opposite role of Mg in the oncology field. Many authors showed that a high content of Mg in the diet is associated with a lower incidence of gastric, colon and breast cancers. However, various data showed that the availability of Mg by cancerous tissues could be involved in the development and/or growth of tumors .

A little is known about the significance of Mg in liver disease. A negative association of primary liver cancer with dietary intake of Mg has been demonstrated .

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old) of both genders with compensated or decompensated liver cirrhosis with or without HCC.

Exclusion Criteria:

* Patients who received Zn or Mg supplementation within the previous 3 months.
* Non-cirrhotic HCC
* Patients with other malignancies.
* Pregnant and lactating women.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults of both genders with compensated or decompensated liver cirrhosis with or without HCC.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Serum levels of Magnesium in cirrhotic patients and HCC | 12 months
  To evaluate the serum level of Magnesium in cirrhotic patients with HCC, and to compare it with the level in cirrhotic patients without HCC and in healthy subjects.
Serum level of Zinc in cirrhotic patients and HCC | 12 months
  To evaluate the serum level of Zinc in cirrhotic patients with HCC, and to compare it with the level in cirrhotic patients without HCC and in healthy subjects.

SECONDARY OUTCOMES:
serum level of Magnesium and the Barcelona clinic classification | 12 months
  To investigate the relationship between serum level of Magnesium and the Barcelona Clinic Liver Cancer (BCLC) stage of HCC.
serum level of Zinc and the Barcelona clinic classification | 12 months
  To investigate the relationship between serum level of Zinc and the Barcelona Clinic Liver Cancer (BCLC) stage of HCC.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al Alawi AM, Majoni SW, Falhammar H. Magnesium and Human Health: Perspectives and Research Directions. Int J Endocrinol. 2018 Apr 16;2018:9041694. doi: 10.1155/2018/9041694. eCollection 2018. PMID 29849626
- [Background] Ferlay J, Colombet M, Soerjomataram I, Parkin DM, Pineros M, Znaor A, Bray F. Cancer statistics for the year 2020: An overview. Int J Cancer. 2021 Apr 5. doi: 10.1002/ijc.33588. Online ahead of print. PMID 33818764
- [Background] Huang WQ, Long WQ, Mo XF, Zhang NQ, Luo H, Lin FY, Huang J, Zhang CX. Direct and indirect associations between dietary magnesium intake and breast cancer risk. Sci Rep. 2019 Apr 8;9(1):5764. doi: 10.1038/s41598-019-42282-y. PMID 30962499
- [Background] Meng Y, Sun J, Yu J, Wang C, Su J. Dietary Intakes of Calcium, Iron, Magnesium, and Potassium Elements and the Risk of Colorectal Cancer: a Meta-Analysis. Biol Trace Elem Res. 2019 Jun;189(2):325-335. doi: 10.1007/s12011-018-1474-z. Epub 2018 Aug 31. PMID 30171595